CLINICAL TRIAL: NCT06072365
Title: Evaluation of the Change in Caloric Intake Before and 12 Months After the Initiation of Treatment With Elexacaftor/Tezacaftor/Ivacaftor, in Patients With Cystic Fibrosis.
Brief Title: Treatment With Elexacaftor/Tezacaftor/Ivacaftor, in Patients With Cystic Fibrosis and Caloric Intake
Acronym: NUTRIMUCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0364; 2021-A02018-33 (Other: ID-RCB)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis
Keywords: caloric intake
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cystic fibrosis: patient with cystic fibrosis treated with With Elexacaftor/Tezacaftor/Ivacaftor,
  Interventions: Other: nutritional intake questionnaire

INTERVENTIONS:
Other: nutritional intake questionnaire — patients completed a nutritional intake questionnaire before to start the treatment, 3mounths after and twelve months after

SUMMARY:
The aim of the study is to describe the evolution of caloric intake in patients with cystic fibrosis with an indication to start treatment with Elexacaftor/Tezacaftor/Ivacaftor according to the Marketing Authorization, between the start of treatment and at 12 months.

DETAILED DESCRIPTION:
Cystic fibrosis is a genetic pathology linked to a dysfunction of the CFTR protein.

Undernutrition is common in the natural course of cystic fibrosis, it is linked to exocrine pancreatic insufficiency but also to the increase in energy expenditure due to respiratory damage.

At a time when these CFTR modulators are greatly modifying the prognosis and management of cystic fibrosis, it is important to describe how caloric and nutritional intake evolve under treatment with Elexacaftor/Tezacaftor/Ivacaftor in order to be able, in the long term, to adapt nutritional recommendations under treatment with CFTR modulators.

The aim of the study is to describe the evolution of caloric intake in patients with cystic fibrosis with an indication to start treatment with Elexacaftor/Tezacaftor/Ivacaftor according to the Marketing Authorization, between the start of treatment and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis
* Patient with an indication to start treatment with Elexacaftor/Tezacaftor/Ivacaftor according to the Marketing Authorization.
* Patient who has not received treatment with CFTR modulators in the 6 months preceding inclusion.
* No opposition expressed by the patient (if ≥ 18 years) or by at least one of the holders of parental authority and the child (if < 18 years).
* Be affiliated to a social security scheme or be a beneficiary of such a scheme.

Exclusion Criteria:

-

Ages: 2 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Refusal to participate
  * Patients and/or holders of parental authority presenting difficulties in understanding and/or communication.
  * Inability to complete a reliable food collection.
  * Any pathological condition making interpretation of results difficult from the investigator's point of view.
  * Transplant patient
  * Pregnant or breastfeeding woman
  * Person under guardianship or curatorship.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
caloric intake 12 months after the beginning of treatment | 12 months
  Describe the evolution of caloric intake in patients with cystic fibrosis with an indication to start treatment with Elexacaftor/Tezacaftor/Ivacaftor according to the Marketing Authorization, between the start of treatment and at 12 months.

SECONDARY OUTCOMES:
caloric intake 3 months after the beginning of treatment | 3 months
  Describe the evolution of caloric intake in patients with cystic fibrosis with an indication to start treatment with Elexacaftor/Tezacaftor/Ivacaftor according to the Marketing Authorization, between the start of treatment and at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marion LAGARRIGUE, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - UHBordeaux, Bordeaux
  - UHLimoges, Limoges
  - UHToulouse, Toulouse

REFERENCES:
- [Derived] Enaud R, Languepin J, Lagarrigue M, Arrouy A, Macey J, Bui S, Dupuis M, Roditis L, Flumian C, Mas E, Mittaine M. Dietary intake remains unchanged while nutritional status improves in children and adults with cystic fibrosis on Elexacaftor/Tezacaftor/Ivacaftor. Clin Nutr. 2025 Jul;50:76-82. doi: 10.1016/j.clnu.2025.04.027. Epub 2025 Apr 30. PMID 40378731